CLINICAL TRIAL: NCT03247595
Title: Efficacy of Magnesium Citrate Capsules in Colonoscopy Preparation: A Randomized, Investigator-blinded Non-inferiority Trial Using Polyethylene Glycol as the Active Control.
Brief Title: Testing How Well Magnesium Citrate Capsules Work as Preparation for a Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1031752
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Colonoscopy
Keywords: Colonoscopy preparation; Magnesium Citrate Capsules
MeSH Terms: interventions — magnesium citrate; polyethylene glycol 3350; Bisacodyl

STUDY DESIGN:
Intervention Model Description: One arm receives Polyethelyne Glycol colonoscopy preparation and the other arm receives magnesium citrate capsules colonoscopy preparation.
Who Masked: Investigator
Masking Description: The endoscopist who reports colon cleanliness is blinded to the subject's assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyethylene Glycol (Active Comparator): Polyethylene Glycol 3350: 4 Liters
  Interventions: Other: Polyethylene Glycol 3350
- Magnesium Citrate Capsules (Experimental): 36 Magnesium citrate capsules
  Interventions: Dietary Supplement: Magnesium Citrate Capsules; Other: Dulcolax Tablets

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate Capsules — 36 magnesium citrate gelatin capsules
  Arms: Magnesium Citrate Capsules
Other: Polyethylene Glycol 3350 — 4 liters of Polyethylene Glycol for colonoscopy preparation
  Arms: Polyethylene Glycol
Other: Dulcolax Tablets — 4 Dulcolox Tablets
  Arms: Magnesium Citrate Capsules

SUMMARY:
This study compares a colonoscopy preparation composed of magnesium citrate capsules to a preparation of polyethylene glycol solution. The hypothesis is that the magnesium citrate capsules work as well and are better liked by patients due to the lack of taste.

ELIGIBILITY:
Inclusion Criteria:

* • Scheduled for colonoscopy at Sinai Hospital or Woodholme GI Associates

Exclusion Criteria:

* • Calculated creatinine clearance under 30ml/min

  * On PPI and unable to stop for five days before colonoscopy
  * On H2 blockers and unable to stop for two days before colonoscopy
  * achlorhydria
  * Previous colon surgery
  * Cardiovascular disease, including uncontrolled congestive heart failure, unstable angina pectoris, or recent (3 months) percutaneous transluminal coronary angioplasty, myocardial infarction, or coronary artery bypass graft surgery
  * Colon disease, including chronic constipation (<2 bowel movements per week for >1 year), ileus and/or acute obstruction, ileostomy, right or transverse colostomy, subtotal colectomy (≥50% of colon removed) with ileosigmoidostomy, hypomotility syndrome, megacolon, or idiopathic pseudo-obstruction
  * Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Colon Cleanliness | During colonoscopy
  Boston scale rating of colon cleanliness

SECONDARY OUTCOMES:
Patient compliance and satisfaction | On the day of colonoscopy
  Patient's experience recorded in a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Dubin, MD, Principal Investigator — LifeBridge Health
Locations (2):
- United States (2):
  - Woodholme Gastroenterology, Baltimore, Maryland
  - Sinai Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rex DK, Johnson DA, Anderson JC, Schoenfeld PS, Burke CA, Inadomi JM; American College of Gastroenterology. American College of Gastroenterology guidelines for colorectal cancer screening 2009 [corrected]. Am J Gastroenterol. 2009 Mar;104(3):739-50. doi: 10.1038/ajg.2009.104. Epub 2009 Feb 24. PMID 19240699
- [Background] Kastenberg D, Barish C, Burack H, Dalke DD, Duckor S, Putnam W, Valenzuela G; INKP-100 Study Group. Tolerability and patient acceptance of sodium phosphate tablets compared with 4-L PEG solution in colon cleansing: combined results of 2 identically designed, randomized, controlled, parallel group, multicenter phase 3 trials. J Clin Gastroenterol. 2007 Jan;41(1):54-61. doi: 10.1097/01.mcg.0000212662.66644.76. PMID 17198066
- [Background] Flemming JA, Vanner SJ, Hookey LC. Split-dose picosulfate, magnesium oxide, and citric acid solution markedly enhances colon cleansing before colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2012 Mar;75(3):537-44. doi: 10.1016/j.gie.2011.09.018. Epub 2011 Dec 21. PMID 22192423
- [Background] Lindberg JS, Zobitz MM, Poindexter JR, Pak CY. Magnesium bioavailability from magnesium citrate and magnesium oxide. J Am Coll Nutr. 1990 Feb;9(1):48-55. doi: 10.1080/07315724.1990.10720349. PMID 2407766
- [Background] Calderwood AH, Schroy PC 3rd, Lieberman DA, Logan JR, Zurfluh M, Jacobson BC. Boston Bowel Preparation Scale scores provide a standardized definition of adequate for describing bowel cleanliness. Gastrointest Endosc. 2014 Aug;80(2):269-76. doi: 10.1016/j.gie.2014.01.031. Epub 2014 Mar 12. PMID 24629422
- [Background] Kastenberg D, Chasen R, Choudhary C, Riff D, Steinberg S, Weiss E, Wruble L. Efficacy and safety of sodium phosphate tablets compared with PEG solution in colon cleansing: two identically designed, randomized, controlled, parallel group, multicenter phase III trials. Gastrointest Endosc. 2001 Dec;54(6):705-13. doi: 10.1067/mge.2001.119733. PMID 11726845